CLINICAL TRIAL: NCT00004579
Title: A Phase I, Dose-Ranging Trial of the Pasteur Merieux Connaught (PMC) Oligomeric HIV-1 gp160MN/LAI-2 Vaccine Alone or Primed With Live Recombinant ALVAC-HIV (vCP205) in HIV Seronegative Adults
Brief Title: A Study to See Whether Two HIV Vaccines Are Safe and Can Prevent HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Prevention
Other Study IDs: RV124
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Vaccines, Synthetic; Viral Vaccines; HIV-1; Dose-Response Relationship, Drug; HIV Envelope Protein gp160; AIDS Vaccines; HIV Seronegativity; Avipoxvirus; Immunization; HIV Envelope Protein gp120; Recombination, Genetic
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: gp160 MN/LAI-2
Biological: ALVAC-HIV MN120TMG (vCP205)

SUMMARY:
The purpose of this study is to see whether an HIV vaccine, ALVAC vCP205, is safe and can prevent HIV infection. The vCP205 vaccine will be tested with another vaccine, gp160MN/LAI-2.

DETAILED DESCRIPTION:
This study consists of 2 parts:

Part A: Dose-escalation protocol using oligomeric gp160MN/LAI-2. Part B: Placebo-controlled, randomized, double-blind (within arm) study of vCP205 priming with gp160MN/LAI-2 boosting.

Volunteers are followed for at least 1 year.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for this study if they:

* Are HIV-negative.
* Are in good health.
* Are between ages 18 and 55.
* Are available for at least 1 year.
* Are a resident of the United States of America.
* Agree to practice sexual abstinence or use birth control.

Exclusion Criteria

Volunteers will not be eligible for this study if they:

* Have ever been given an HIV vaccine or certain other vaccines. (However, rabies vaccines are allowed.)
* Participate in activities that place them at high-risk for HIV infection, such as injection drug use or unprotected sex with someone who has HIV infection.
* Have certain psychiatric, medical, or substance abuse problems.
* Are allergic to eggs or other vaccines.
* Are an employee at a participating site and have access to study information.
* Are taking certain medications.
* Have received blood transfusions within 3 months before entering this study.
* Are pregnant or breast-feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 1998-04

CONTACTS AND LOCATIONS:
Overall Officials: Jerome H. Kim, Principal Investigator
Locations (1):
- Walter Reed Army Institute of Research, Rockville, Maryland, United States

REFERENCES:
- [Background] Kim J, Robb M, Cox J, Ratto-Kim S, Vancott T, Zahwa H, Malia J, Chaddic C, El Habib R, Caudrelier P, Klein M, Excler JL, Birx D, McNeil J. Humoral and cellular HIV-specific responses induced by the prime-boost combination of Aventis-Pasteur ALVAC-HIV (vCP205) and oligomeric HIV-1 gp160MN/LAI-2 in HIV-uninfected adults. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 179)
- [Derived] O'Connell RJ, Excler JL, Polonis VR, Ratto-Kim S, Cox J, Jagodzinski LL, Liu M, Wieczorek L, McNeil JG, El-Habib R, Michael NL, Gilliam BL, Paris R, VanCott TC, Tomaras GD, Birx DL, Robb ML, Kim JH. Safety and Immunogenicity of a Randomized Phase 1 Prime-Boost Trial With ALVAC-HIV (vCP205) and Oligomeric Glycoprotein 160 From HIV-1 Strains MN and LAI-2 Adjuvanted in Alum or Polyphosphazene. J Infect Dis. 2016 Jun 15;213(12):1946-54. doi: 10.1093/infdis/jiw059. Epub 2016 Feb 11. PMID 26908741